CLINICAL TRIAL: NCT03118401
Title: Stool Ritual: Impact on the Number of Nights Without Stools Among Dependent Residents in Institutions for Dependent Elderly People
Acronym: RITUELIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I16025 (RITUELIM)
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Homes for the Aged; Intestinal Elimination

STUDY DESIGN:
Intervention Model Description: At the end of the first 4 weeks of collection of the data on an individual stool diary with usual care of the resident, a randomization will be carried out dividing the patients according to the following groups:
  1. / Experimental group Implementation period: From the stool diary: - determine the stool profile of each resident over 1 week (W5)
  2. / Control group: without modification of practices and without data collection from W5 to W6.
  At the end of this second period, data were collected on an individual stool diary in each of the two groups for 4 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ritual of stool (Experimental): During the first 4 weeks, data will be collected on an individual stool diary with usual care of the resident After randomization will start the implementation period of ritual of stool. From the stool diary: - will be determined the stool profile of each resident over 1 week and application of the ritual of stool the following week At the end of this second period, data will be collected on an individual stool diary in for 4 weeks
  Interventions: Other: Ritual of stool
- Usual practice (Other): During the first 4 weeks, data will be collected on an individual stool diary with usual care of the resident After randomization will start 2 weeks without data collection. Patient will be follow in usual practice.
  At the end of this second period, data will be collected on an individual stool diary in for 4 weeks
  Interventions: Other: Usual practice

INTERVENTIONS:
Other: Ritual of stool — During the first 4 weeks, data will be collected on an individual stool diary with usual care of the resident After randomization will start the implementation period of ritual of stool. From the stool diary: - will be determined the stool profile of each resident over 1 week and application of the ritual of stool the following week At the end of this second period, data will be collected on an individual stool diary in for 4 weeks
  Arms: Ritual of stool
Other: Usual practice — During the first 4 weeks, data will be collected on an individual stool diary with usual care of the resident After randomization will start 2 weeks without data collection. Patient will be follow in usual practice.
  At the end of this second period, data will be collected on an individual stool diary in for 4 weeks
  Arms: Usual practice

SUMMARY:
As they age, the intestinal elimination function can be altered by external factors. Sleeping is also a vital need for maintaining health. Sleep time varies with age (from 18h / day for an infant to 7h30 on average for an adult) and sleep disorders increase with age (INSERM source). In our study, the night is from 9 pm to 7 am, corresponding to the working hours of the night shift. Between 42% and 50% of episodes of wakefulness of more than 4 minutes in EHPAD are due to noise, light or the practice of care related to incontinence. 87% of all incontinence care practices have been associated with wake-up episodes. A personalized day care program would allow residents to improve the quality of their sleep by minimizing stools at night and therefore interventions by caregivers.

The ritual of stools, can be defined as the set of rules to observe to defecate in good physiological, physical conditions:

* Be in a suitable place for intestinal elimination: personal bathroom preferably on the toilet or on a pierced chair that will perhaps be more secure and comfortable with the armrests. The position to be taken is important.
* Propose a small bench to put under the feet to raise the knees higher than the hips and increase the abdominal pressure.
* Preserve the visual and auditory intimacy of the resident at the time of defecation. Failure to do so may result in the person repressing his desire to defecate.
* Allow the resident the time needed on the toilets the doorbell at hand and with the assurance that the caregiver will come back in a short time. Do not press it and do not forget it, privilege the autonomy and check that there is toilet paper.

The establishment of the stool ritual is not intended to reduce the amount of stool by day, but it aims to postpone the nighttime exemption on the day, and does not prevent the stool emission to other times of the day or night.

ELIGIBILITY:
Inclusion Criteria:

* Dependent elderly people living in institutions for elderly dependents.
* GIR 1 or 2
* Residents being able to sit in a seated position on a pierced chair or a safe toilet.
* Residents who have lived in the institution for at least 1 month in order to limit the biases due to the change of place of life

Exclusion Criteria:

* Residents with the physical and cognitive abilities to go to the toilet alone wisely.
* Residents with stomies
* Residents with a history of intestinal occlusion
* Residents participating in another study.
* Residents under guardianship or safeguard justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Number of nights with stools during the follow-up period | Week 10
  Number of nights with stools during the follow-up period

SECONDARY OUTCOMES:
Evolution in number of nights with stool | Week 10
  Difference in number of nights with stool between initial observation period and follow-up period in each of the 2 randomization groups
Evolution in number of laxative medication | Week 10
  Difference in the number of laxative medication between initial observation period and follow-up period in each of the 2 randomization groups
Satisfaction questionary | Week 10
  At the end of the study, satisfaction of the caregivers who participated in the implementation of the ritual of stools concerning the interest of this ritual by means of a satisfaction questionary

CONTACTS AND LOCATIONS:
Overall Officials: Pascale SEIGNEURIN-HERISSE, Principal Investigator — Ussel Hospital
Locations (1):
- EHPAD les Ecureuils, Ussel, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Seigneurin-Herisse P, Toniolo J, Marchat N, Micallef L, Labrunie A, Delaide V, Beloni P. Impact of a person-centered bowel program on the frequency of nights with bowel movement in dependent elderly people in nursing home: A single-centre randomized controlled trial. Int J Nurs Stud. 2022 Nov;135:104348. doi: 10.1016/j.ijnurstu.2022.104348. Epub 2022 Aug 13. PMID 36088731